CLINICAL TRIAL: NCT00001125
Title: Use of a Live-Attenuated Varicella-Zoster Virus (VZV) Vaccine to Boost Immunity to VZV in HIV-Infected Children Previously Infected With Varicella
Brief Title: Use of a Varicella-Zoster Virus (VZV) Vaccine to Prevent Shingles in HIV-Infected Children Who Have Already Had Chickenpox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: PACTG 391; 10614 (Registry Identifier: DAIDS ES Registry Number); ACTG 391
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Chickenpox
Keywords: Antibodies, Viral; Chickenpox; Chickenpox Vaccine
MeSH Terms: conditions — HIV Infections; Chickenpox | interventions — Herpes Zoster Vaccine

INTERVENTIONS:
Biological: Varicella Virus Vaccine (Live)

SUMMARY:
The purpose of this study is to see if the varicella-zoster virus (VZV) vaccine will be safe and if it can help prevent shingles in HIV-infected children who have already had chickenpox.

VZV is the virus that causes chickenpox. If this virus is reactivated in the body, it can also cause shingles. Shingles is common in children with HIV who have had chickenpox, although it is usually not life-threatening. The VZV vaccine used in this study may be able to prevent HIV-positive children who have had chickenpox from developing shingles.

DETAILED DESCRIPTION:
Varicella (chickenpox) results from primary infection with VZV. Varicella, a common and usually benign illness in normal children, is more severe in HIV-infected children and may result in other conditions such as HZ (shingles). HZ is due to reactivation of latent VZV acquired during varicella and is common in HIV-infected children who have had natural varicella. While HZ is not likely to be life-threatening in these children, it does cause considerable morbidity and interferes with quality of life. Use of a live-attenuated VZV vaccine may be able to boost immunity in these children.

Two immunologic cohorts are enrolled. Cohort A includes children with a CD4 cell percentage greater than or equal to 20 percent that has been documented as stable for at least the 6 months prior to the time varicella developed (confirmed by a minimum of 2 tests) and a CD4 cell percentage greater than [AS PER AMENDMENT 10/27/99: or equal to] 15 percent that has been documented as stable for at least the 6 months prior to enrollment (confirmed by a minimum of 2 tests). Cohort B includes children with a CD4 cell percentage greater than or equal to 10 percent and less than 15 percent that has been documented as stable for at least the 6 months prior to the time varicella developed and stable for at least the 6 months prior to enrollment (confirmed by a minimum of 2 tests). [AS PER AMENDMENT 4/20/01: Cohort B includes children who have a CD4 cell percentage less than 15% documented by a minimum of 1 but preferably 2 tests within 1 year of onset of varicella (i.e., within 1 year before to 1 year after varicella) and a CD4 cell percentage greater than or equal to 15% documented by a minimum of 2 tests at the time of enrollment.] A pilot study precedes the full study. [AS PER AMENDMENT 10/27/99: The pilot study for Cohort A precedes the full study for Cohort A and the pilot study for Cohort B. The pilot study for Cohort B precedes the full study for Cohort B.] The pilot study includes 10 children from each cohort who receive live-attenuated VZV at Weeks 0 and 8. If 3 pilot-study patients in a cohort meet a toxicity endpoint related to the vaccine, the dose regimen has failed the safety criteria for that cohort. [AS PER AMENDMENT 10/27/99: If 3 children in the pilot study for Cohort A meet a toxicity endpoint deemed to be related to the vaccine, the dose regimen has failed safety criteria for both cohorts. If 3 children in the pilot phase of Cohort B meet a toxicity endpoint deemed related to the vaccine, the dose regimen has failed the safety criteria for Cohort B.] If, at 12 weeks after immunization, at least 5 pilot-study patients in a cohort respond and the safety profile is deemed adequate, the pilot study extends into a full study with the immunization of an additional 20 patients from that cohort. [AS PER AMENDMENT 10/27/99: If, at Week 12, at least 5 pilot-study patients in Cohort A meet immunologic criteria and the safety profile is deemed adequate, then the full study for Cohort A and the pilot study for Cohort B opens. If the same immunologic and safety criteria are met for the pilot study for Cohort B, then the full study for Cohort B opens.] If either cohort shows an inadequate immunologic response or safety profile, the study team reviews the results to determine if another regimen should be considered. In the full study, patients receive 2 immunizations, at Weeks 0 and 8. Varicella antibody titers and in vitro responder cell frequency (RCF) assays are measured at Weeks 0, 4, 8, 12, 24, 52, 78, and 104. Symptoms, HIV progression, and VZV presence are monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are 2 to 18 years old (need consent of parent or guardian if under 18).
* Are HIV-positive.
* Are VZV-positive.
* Have a CD4 cell percentage of at least 15 percent at the time of enrollment. (This criterion reflects a change from the original CD4 cell percentage.)
* Have been receiving stable anti-HIV therapy for at least 3 months, with no plans to change these medications.
* Had chickenpox at least 6 months prior to study entry.
* Were at least 1 year old when they had chickenpox.
* Agree to use a barrier method of birth control (such as a condom) during the study.

Exclusion Criteria

Children will not be eligible for this study if they:

* Have an active infection within 72 hours of study entry.
* Have a fever over 101 F within 72 hours of study entry.
* Were exposed to chickenpox or shingles within 4 weeks prior to study entry.
* Have ever had shingles.
* Live with someone who has HIV, or who has a weak immune system, and has never had chickenpox.
* Have taken certain medications that affect the immune system, such as steroids, within 30 days of study entry.
* Have taken or are planning to take VZIG or IVIG within 1 year prior to or 2 months after a study vaccination.
* Are allergic to the vaccine, or to neomycin.
* Have received or expect to receive another vaccine within 30 days prior to or 30 days after a study vaccination.
* Have ever received a chickenpox vaccine.
* Are taking aspirin or expect to use aspirin 6 weeks after a study vaccination.
* Have taken or plan to take any anti-herpes drugs within 1 week before or 3 weeks after a study vaccination.
* Have received or plan to receive a blood transfusion within 1 year before or 2 months after a study vaccination.
* Have certain medical problems that would interfere with the study.
* Are pregnant or breast-feeding.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Gershon, Study Chair
Locations (22):
- United States (22):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - Cooper Univ. Hosp., Camden, New Jersey
  - NJ Med. School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Cornell Univ., Div. of Ped. Infectious Diseases & Immunology, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Vanderbilt Univ. Med. Ctr., Div. of Ped. Infectious Diseases, Nashville, Tennessee